CLINICAL TRIAL: NCT06986122
Title: Controllability of Virtual Contexts for the Modulation of the Affective Experience
Brief Title: Virtual Contexts for Affective Modulation
Acronym: VCAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor in Neuroscience, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00033386
Record Dates: First submitted 2025-05-08; First posted 2025-05-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pain Control; Anxiety; Memory
Keywords: Place conditioning; controllability of pain
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contextual learning (Experimental): All participants complete trials in three virtual contexts (safe, controllable threat, uncontrollable threat), with pain controllability and task performance assessed across all conditions in a randomized within-subject design.
  Interventions: Behavioral: Pain Threat Manipulation; Behavioral: Pain Controllability Manipulation

INTERVENTIONS:
Behavioral: Pain Threat Manipulation — Participants receive brief thermal pain stimuli in certain virtual environments to examine how threat influences perception and physiological responses.
Behavioral: Pain Controllability Manipulation — In some contexts, participants can reduce or avoid pain using a button; in others, no action changes the outcome. This manipulation is used to study the effects of perceived control over pain.

SUMMARY:
This study investigates how spatial context and perceived controllability modulate pain, affective states such as anxiety, and motivated behavior. The study examines how control over pain and threat-related environments influences pain perception, state anxiety, associated autonomic responses, and behavior. The main questions it aims to answer are:

Does having control over pain within specific contexts alter how much pain people feel-even when the stimulus intensity remains constant? How do different types of environments (safe, controllable, or uncontrollable) shape pain-related brain activity, subjective anxiety, and physiological arousal? How do people perform cognitively demanding or distracting tasks (and retain their memory) when under threat versus when in control? Lastly, how do these learned associations with spatial contexts persist or adapt when environmental contingencies are explicitly changed?

Taken together, exploration of these factors may lay the groundwork for understanding how placebo-related mechanisms-including perceived control, contextual learning, emotional engagement, and distraction-interact to shape pain and anxiety in complex environments.

DETAILED DESCRIPTION:
The study investigates how perceived controllability and threat-related spatial contexts influence pain perception, affective state, autonomic responses, and behavior. Specifically, it aims to dissect the systems-level mechanisms by which humans interpret and respond to painful experiences in environments that differ in perceived threat and agency. These mechanisms-spanning from pain perception to context-driven learning and flexible adaptation-are central to understanding both everyday coping and the cognitive underpinnings of placebo effects.

Participants will explore three distinct virtual rooms, each associated with a different contingency: one room is safe (no pain), one involves controllable threat (participants can use a button to temporarily suppress incoming thermal pain), and one involves uncontrollable threat (pain occurs and cannot be avoided). The context-pain contingencies are learned across repeated exposures. While in each room, participants will also engage in a distracting maze-navigation task requiring them to press a sequence of levers to escape. This setup allows measuring immediate control over pain (via the button) and motivated behavior under threat (via navigation performance).

Following primary outcomes are measured:

1. Subjective pain reports following each stimulus,
2. Anxiety responses (based on self-reports and inferred from autonomic responses e.g., skin conductance, breathing, heart rate).

In addition, navigation behavior and brain activity via functional MRI is also monitored (as subjects perform various tasks inside the scanner).

In a later phase, extinction or reversal learning will occur: all rooms will deliver identical, uncontrollable pain, or participants will be instructed that previous contingencies have changed. Here the investigators probe how learned threat and control associations persist, generalize, or adapt, and how placebo-relevant mechanisms like expectation, context, and cognitive reappraisal interact to shape pain and behavior. By independently manipulating context, control, and task goals, this design captures a rich profile of how humans flexibly regulate threat and pain in complex environments. This is a key step in examining the key factors that may contribute to the placebo effect under a joint paradigm: namely, the agency/controllability, place context and engagement/distraction.

The following aims are examined in this study:

Aim 1: How spatial contexts associated with safety, controllable threat, or uncontrollable threat influence subjective pain perception and behavioral responses. The first hypothesis is that controllability of pain (Context B vs C) could produce analgesia. This controllability associated with context is likely to persist during extinction.

Aim 2: The investigators aim to characterize the neural circuits supporting contextual threat learning, controllability, and pain modulation. The second hypothesis is that the hippocampus will differentiate spatial contexts, Amygdala will show heightened activity in the uncontrollable threat context, and analgesia may incorporate activity in periaqueductal gray (PAG) and opioid-related midbrain circuits.

Aim 3: The third aim is to examine the effect of threat and behavioral control on the autonomic markers such as breathing, skin-conductance and heart rate. The corresponding hypothesis is that a multidimensional marker of threat-state and anxiety could be derived from these features that may be sensitive to various contexts and controllability.

Aim 4: Next aim is to study how the affective state induced by different threat contexts (safe, controllable, uncontrollable) modulates incidental visual memory for the contexts.

Aim 5: The final is aim to study how the context-outcome associations are generalized to new contexts and dynamically updated when subjects are explicitly instructed to do so. The corresponding hypothesis is that this generalization or reversal might be dependent upon hippocampus-OFC interactions.

The study design consists of the following sessions:

1. Session 1: Consent, Familiarization, and Baseline Assessment (~1.5 hours):

   As part of the screening process, a pain calibration procedure is performed on each participant in order to ensure that all temperatures delivered during any subsequent procedures are within participants' tolerable range. The pain calibration procedure consists of applying a range of temperatures to various sites on the subject's skin. Participants rate each stimulus using the provided scale and respond to two prompts ("Painful?" and "Tolerable?"). The ratings are used to fit a mathematical relationship between noxious stimulus and reported pain. Subjects will not be permitted to continue participation if their pain tolerances are too high (hypersensitive) or too low (hyposensitive) -i.e., those that would require delivery of temperatures above the boundaries stipulated by the guidelines in this protocol, or that do not allow for sufficient experimental variation of the temperatures delivered.

   Further, subjects will be familiarized with virtual contexts without any pain. Participants will explore 3 visually distinct virtual "rooms" (contexts A, B, C) via a non-immersive VR setup (e.g., monitor-based navigation). Participants learn to recognize rooms but are not told of any contingencies. Participants navigate through the rooms in a block of 15 trials (5 trials per context, 1 trial ≈ 1-1.5 min) and learn to solve an escape task (by activating a set of levers in a sequence). Subjects are later tested on a spatial context identification task to confirm room encoding (with participants performing below chance removed from the study).
2. Session 2: Threat Learning and Controllability Manipulation (~1 hour):

   The experimental session will be conducted in the MRI. Following a consenting process, participants will be acquainted with MRI safety guidelines. Once in the scanner, subjects will perform the task in 4 blocks of 15 trials each (60 trials, 1 trial = 1-2 minutes, 20 trials per context). In each room, subjects learn to perform a navigational task (such as activating a sequence of switches) to proceed to the next room.

   Each virtual room is paired with consistent contingency. Room A: Safe - no pain is delivered. Room B: Controllable threat - pain is delivered but can be avoided by pressing a button that the subjects have access to.

   Room C: Uncontrollable threat - pain is delivered and cannot be avoided (statistically similar amount of pain is administered as Room B).

   In each trial, participants rate pain, perceived control, and room aversiveness. Subjects' autonomic responses and behavioral responses (e.g. instantaneous position, velocity etc.) are recorded throughout the sessions. A T1 anatomical image of the subject's brain will also be acquired to localize the ROIs.

   Following the training, subjects perform a visual memory task where they are shown images from the three contexts as well as novel ones and asked to report if they recall seeing them.
3. Session 3: Extinction (~1.5-2 hours) In the subsequent session, all three rooms are now presented with uncontrollable pain, regardless of prior association. Participants are not informed of the change; the goal is to assess spontaneous extinction and memory persistence. The session has the same trial timing and structure as Session 2.
4. Session 4-5: Reversal and generalization blocks (~1.5-2 hours) For a subset of subjects, after initial extinction, the threat conditions are reinstated. Following the reinstatement, the contingencies are reversed (e.g., Room B now becomes unsafe). Participants are explicitly instructed about the reversal (instructed learning). The remaining trial structure is similar to session-2. Subjects are also presented with novel contexts that may be similar or dissimilar to the original contexts.

Before each session, participants are advised to get 8 hours of sleep, and not to consume any alcohol or central acting drugs or pain medication for at least 24 h before each experiment.

Below are the set of detailed hypotheses for the study:

1. Pain Report: Pain is lower in controllable context (B) than uncontrollable (C) in Session 2; in Session 3, pain reports will reflect memory of control: B < C > A, even though all contexts are now uncontrollable.
2. Autonomic Arousal: Skin conductance and breathing rate can distinguish C vs. A (threat vs. safety); threat signals will be lower in B than C during Session 2, and in Session 3, threat memory will persist: C > B > A. Similarly, self-reported anxiety will be higher in the uncontrollable context (C) than in B or A, and may correlate with autonomic arousal.
3. Pain Report + Autonomic: Individuals showing stronger autonomic arousal in C will also report higher pain, even with identical stimulation.
4. Navigational Efficiency: Task performance may differ between B and C due to the cognitive load of controlling pain under threat.
5. Incidental Visual Memory: Memory for visual details may be enhanced in high-arousal contexts (C).

Together, this multi-session design provides a comprehensive framework to investigate how controllability, spatial context, and cognitive engagement interact to shape pain, anxiety, and adaptive behavior. The findings from the study form a foundation for understanding placebo-like modulation of pain and affect in complex, real-world environments.

ELIGIBILITY:
* No self-reported current or history of depression, bipolar disorder, or other psychiatric diagnosis
* No self-reported current seizure disorder (i.e., seizure within past 10 years), or history of stroke or other major neurological diagnosis
* No self-reported current chronic pain, or acute pain within three months of the study period
* No current migraine disorder (i.e., 15 headache days or more in 1 month)
* No use of central nervous system-effective medication or other medication for neurological/psychiatric treatment
* No self-reported substance abuse within the last six months
* No contraindication to MRI (e.g., pregnancy, claustrophobia, pacemakers, ear/cochlear implants, shrapnel injuries, clips, or other ferromagnetic/electrical objects/devices, diagnosed brain abnormality such as tumor, or skin lesions on the scalp.)
* No contraindications for induced pain (e.g., no heart disease, high blood pressure, heart surgery, heart problems of any kind, severe asthma, respiratory problems of any kind, fibromyalgia, Raynaud's Syndrome or Disease, chronic pain, diabetes)
* Participants must be capable of performing experimental tasks (e.g., are able to read), are fluent or native speakers of English
* Participants must be able to tolerate the maximum level of thermal pain stimuli (for thermal stimuli)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Ratings | 3-10 sec post-stimulus throughout testing sessions, on average complete within 1 month
  Self-reported pain level following each thermal stimulus, measured on a visual analog scale. 0-100 scale with 0 indicating no pain and higher values indicating more pain.
Self-Reported Anxiety Ratings | Every 45-60 sec throughout testing sessions, on average complete within 1 month
  Participants rate their current level of anxiety using a 0-100 visual analogue Subjective Units of Distress Scale (SUDS). 0 indicates no anxiety and higher values indicating more anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared to assist with any supplementary or meta-analyses after de-identification of subjects.

REFERENCES:
- [Background] Tzschentke TM. Measuring reward with the conditioned place preference paradigm: a comprehensive review of drug effects, recent progress and new issues. Prog Neurobiol. 1998 Dec;56(6):613-72. doi: 10.1016/s0301-0082(98)00060-4. PMID 9871940
- [Background] Salomons TV, Nusslock R, Detloff A, Johnstone T, Davidson RJ. Neural emotion regulation circuitry underlying anxiolytic effects of perceived control over pain. J Cogn Neurosci. 2015 Feb;27(2):222-33. doi: 10.1162/jocn_a_00702. PMID 25208742
- [Background] Salomons TV, Johnstone T, Backonja MM, Davidson RJ. Perceived controllability modulates the neural response to pain. J Neurosci. 2004 Aug 11;24(32):7199-203. doi: 10.1523/JNEUROSCI.1315-04.2004. PMID 15306654
- [Background] Kragel PA, Kano M, Van Oudenhove L, Ly HG, Dupont P, Rubio A, Delon-Martin C, Bonaz BL, Manuck SB, Gianaros PJ, Ceko M, Reynolds Losin EA, Woo CW, Nichols TE, Wager TD. Generalizable representations of pain, cognitive control, and negative emotion in medial frontal cortex. Nat Neurosci. 2018 Feb;21(2):283-289. doi: 10.1038/s41593-017-0051-7. Epub 2018 Jan 1. PMID 29292378
- [Background] Atlas LY, Bolger N, Lindquist MA, Wager TD. Brain mediators of predictive cue effects on perceived pain. J Neurosci. 2010 Sep 29;30(39):12964-77. doi: 10.1523/JNEUROSCI.0057-10.2010. PMID 20881115
- [Background] Amat J, Baratta MV, Paul E, Bland ST, Watkins LR, Maier SF. Medial prefrontal cortex determines how stressor controllability affects behavior and dorsal raphe nucleus. Nat Neurosci. 2005 Mar;8(3):365-71. doi: 10.1038/nn1399. Epub 2005 Feb 6. PMID 15696163
- [Background] Alvarez RP, Biggs A, Chen G, Pine DS, Grillon C. Contextual fear conditioning in humans: cortical-hippocampal and amygdala contributions. J Neurosci. 2008 Jun 11;28(24):6211-9. doi: 10.1523/JNEUROSCI.1246-08.2008. PMID 18550763